CLINICAL TRIAL: NCT02946203
Title: Prospective Comparison of VoLumen and Breeza Oral Contrast Agents in Pediatric Patients Undergoing CT and MR Enterography
Brief Title: Comparison of VoLumen and Breeza Oral Contrast Agents in Pediatric Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: CIN_Breeza_001
Record Dates: First submitted 2016-10-04; First posted 2016-10-27 (Estimated); Last update posted 2018-02-13 (Actual); Status verified 2018-02

CONDITIONS: Inflammatory Bowel Diseases
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — Barium Sulfate

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Flavored Beverage Oral Contrast-Breeza (Active Comparator): Pediatric patients that are undergoing awake CT and MR enterography at the Cincinnati Children's Hospital Medical Center (CCHMC) base (Burnett) campus will be randomized to either VoLumen (current standard of care oral contrast) or Breeza.
  Interventions: Other: Flavored beverage Oral Contrast
- Barium Sulfate Oral Contrast-VoLumen (Active Comparator): Pediatric patients that are undergoing awake CT and MR enterography at the CCHMC base (Burnett) campus will be randomized to either VoLumen (current standard of care oral contrast) or Breeza.
  Interventions: Other: Barium Sulfate

INTERVENTIONS:
Other: Barium Sulfate — Barium Sulfate Oral Contrast-VoLumen
  Other Names: VoLumen
  Arms: Barium Sulfate Oral Contrast-VoLumen
Other: Flavored beverage Oral Contrast — Flavored beverage for neutral abdominal/pelvic imaging
  Other Names: Breeza
  Arms: Flavored Beverage Oral Contrast-Breeza

SUMMARY:
In this research study, two different oral contrast materials that can be used for CT or MR enterography will be studied. This study is designed to compare which oral contrast material (VoLumen or Breeza) is preferred by pediatric patients and which provides higher quality exams.

DETAILED DESCRIPTION:
VoLumen, a low Hounsfield unit 0.1% barium sulfate suspension that also contains sorbitol and a gum, is the most common oral contrast material used in children and adults undergoing CT and MR enterography (advanced imaging tests used to evaluate the bowel lumen and bowel wall in children and adults, usually with suspected or known Crohn disease). This contrast material is typically administered orally to non-sedated patients during the 45-60 minute period prior to imaging. The goal of oral contrast material administration is to completely fill the small bowel with fluid at the time of imaging. Benefits of oral contrast material at cross-sectional enterography include: improved delineation of bowel from non-bowel structures in the abdomen and pelvis, improved accuracy when assessing bowel wall thickness, and improved visualization of mucosal hyper-enhancement in the setting of active intestinal inflammation.

In some children (and adults), the standard-of-care contrast agent (VoLumen) is poorly tolerated. This is likely due to a variety of factors, including taste, texture, and the volume that is required to be consumed. Recently, a new oral contrast material called "Breeza for neutral abdominopelvic imaging" (or simply Breeza) has become available for use at CT and MR enterography. This agent contains sorbitol, mannitol, and xantham gum (a thickening agent), and it is marketed as a "flavored beverage" as it contains no active ingredient (e.g., barium sulfate). A single study performed in adult volunteers has shown that this new agent performs similar to VoLumen, has a superior taste, and is associated with greater willingness for repeat drinking.

The objective of our study is to compare our standard-of-care oral contrast material to the newly available contrast material in a prospective, randomized, blinded manner. Primary outcomes will include degree of small bowel opacification, distention of the terminal ileum, and patient acceptance/tolerability.

ELIGIBILITY:
Inclusion Criteria:

* Age > 8 years and < 18 years
* Patients undergoing clinically indicated CT or MR enterography

Exclusion Criteria:

* Age < 8 years and ≥ 18 years
* Requirement for sedation for CT or MRI enterography
* Cannot drink oral contrast (will require tube administration)

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 66 (Actual)
Dates: Start 2016-11; Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Degree of bowel opacification as determined by estimated percentage of overall small bowel opacification | 1 year
  To compare the degree of bowel opacification provided by Breeza vs. VoLumen oral contrast materials in pediatric patients undergoing CT and MR enterography. The degree of bowel opacification will be rated 0-100 percent.
Degree of bowel opacification, rated subjectively as excellent, diagnostic, suboptimal or poor | 1 year
  To compare the degree of bowel opacification provided by Breeza vs. VoLumen oral contrast materials in pediatric patients undergoing CT and MR enterography.
Degree of bowel distention as determined by measurement of the largest diameter, normal, small bowel loop in each of the four abdominal quadrants | 1 year
  To compare the degree of bowel distention, measured in millimeters, provided by Breeza vs. VoLumen oral contrast materials in pediatric patients undergoing CT and MR enterography
Degree of bowel distention rated subjectively as excellent, diagnostic, suboptimal or poor | 1 year
  To compare the degree of bowel distention provided by Breeza vs. VoLumen oral contrast materials in pediatric patients undergoing CT and MR enterography

SECONDARY OUTCOMES:
Tolerability as assessed by patient survey with respect to overall tolerability, taste and texture | 1 year
  To compare the patient tolerability of Breeza vs. VoLumen oral contrast materials in pediatric patients undergoing CT and MR enterography as assessed by patient survey using the Likert scale rating of 0-10
Tolerability as assessed by patient survey with respect to abdominal symptoms as well as overall state of well-being | 1 year
  To compare the patient tolerability of Breeza vs. VoLumen oral contrast materials in pediatric patients undergoing CT and MR enterography as assesses by patient survey using the Likert scale rating of 0-10

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Dillman, MD, MSc, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dillman JR, Adler J, Zimmermann EM, Strouse PJ. CT enterography of pediatric Crohn disease. Pediatr Radiol. 2010 Jan;40(1):97-105. doi: 10.1007/s00247-009-1465-5. Epub 2009 Nov 20. PMID 19936733
- [Background] Mollard BJ, Smith EA, Dillman JR. Pediatric MR enterography: technique and approach to interpretation-how we do it. Radiology. 2015 Jan;274(1):29-43. doi: 10.1148/radiol.14122449. PMID 25531478
- [Background] Towbin AJ, Sullivan J, Denson LA, Wallihan DB, Podberesky DJ. CT and MR enterography in children and adolescents with inflammatory bowel disease. Radiographics. 2013 Nov-Dec;33(7):1843-60. doi: 10.1148/rg.337105140. PMID 24224581
- [Background] Young BM, Fletcher JG, Booya F, Paulsen S, Fidler J, Johnson CD, Huprich J, Barlow J, Trout A. Head-to-head comparison of oral contrast agents for cross-sectional enterography: small bowel distention, timing, and side effects. J Comput Assist Tomogr. 2008 Jan-Feb;32(1):32-8. doi: 10.1097/RCT.0b013e318061961d. PMID 18303285
- [Background] Absah I, Bruining DH, Matsumoto JM, Weisbrod AJ, Fletcher JG, Fidler JL, Faubion WA Jr. MR enterography in pediatric inflammatory bowel disease: retrospective assessment of patient tolerance, image quality, and initial performance estimates. AJR Am J Roentgenol. 2012 Sep;199(3):W367-75. doi: 10.2214/AJR.11.8363. PMID 22915428
- [Background] Kolbe AB, Fletcher JG, Froemming AT, Sheedy SP, Koo CW, Pundi K, Bruining DH, Tung J, Harmsen WS, Barlow JM, Fidler JL. Evaluation of Patient Tolerance and Small-Bowel Distention With a New Small-Bowel Distending Agent for Enterography. AJR Am J Roentgenol. 2016 May;206(5):994-1002. doi: 10.2214/AJR.15.15260. Epub 2016 Mar 21. PMID 26998661